CLINICAL TRIAL: NCT06510322
Title: Sildenafil to Reduce Vascular Remodeling During Left Ventricular Assist Device Support
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-16098; 1R01HL172972 (NIH)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sildenafil (Active Comparator): Participants in this arm will receive sildenafil 20mg every 8 hours for 1 week and then dose will be up titrated to 40mg every 8 hours for the duration of the study period.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Participants in this arm will receive matching placebo, which serves as a negative control to understand changes in small and large blood vessels.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Orally administered phosphodiesterase-5 (PDE-5) inhibitor, which enhances nitric oxide signaling in platelets and blood vessels.
  Arms: Sildenafil
Other: Placebo — Matched capsule not containing any medication
  Arms: Placebo

SUMMARY:
Contemporary left ventricular assist device (LVAD) therapy improves survival during advanced heart failure but vascular aging develops rapidly leading to major adverse events including stroke and bleeding in nearly half of patients. In this study, the study team aims to investigate whether sildenafil pharmacotherapy, which has anti-fibrotic effects, can reduce vascular aging during LVAD support. An aim of this study is to compare changes in small blood vessels in the gastrointestinal tract between participants receiving sildenafil or placebo. Video capsule endoscopy (VCE) will be used to assess these changes in small blood vessels.

DETAILED DESCRIPTION:
Over 6.5 million individuals in the United States suffer from heart failure (HF), with the burden of this disease expected to grow over the next decade. Approximately 300,000 of these patients have advanced HF and may benefit from durable left ventricular assist device (LVAD) therapy, which can improve outcomes during advanced HF. However, despite advancements in device design that have increased survival rates, large registries of real- world cases reveal that nearly half of patients experience severe vascular adverse events, including stroke and bleeding, during prolonged contemporary LVAD support. This elevated adverse-event rate remains a major barrier to safely expanding the use and durability of LVAD therapy. Vascular remodeling or aging of the large and small blood vessels is known to promote stroke and bleeding within the general population. Critically, such remodeling is rapidly accelerated under conditions of reduced pulsatility produced by LVADs, evidenced by large vessel stiffening and fibrosis, small vessel angiodysplasia, and endothelial dysfunction. Phosphodiesterase-5 inhibitors (PDE5i), such as sildenafil, are prescribed to select LVAD patients with pulmonary hypertension and right heart failure. However, given that these agents enhance nitric oxide-cGMP signaling in platelets and vascular smooth muscle cells, leading to anti-thrombotic and anti-fibrotic effects, they may also reduce vascular remodeling and related adverse events. Here, based on preliminary findings, a double-blind, randomized, placebo-controlled trial will be conducted to determine the effects of chronic sildenafil administration on vascular remodeling during LVAD support.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Supported by a durable LVAD or planned to undergo placement of a durable LVAD
* Be able to give informed consent

Exclusion Criteria:

* History of pre-existing aortic valve prosthesis or an aortic graft
* Allergy to sildenafil
* Taking any nitric oxide (NO) donor medications
* History of complete carotid occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Aortic Pulse Wave Velocity | From Baseline to 180 days
  Pulse wave velocity (PWV) will be measured by vascular ultrasound. PWV will be calculated by dividing the distance between the carotid and femoral artery waveform acquisition sites (in meters) by the carotid-femoral transit time (change in time, in seconds). Change in group mean PWV from baseline will be summarized. Increases in PWV can be an indicator of vascular fibrosis and are associated with increased risk of cardiovascular comorbidities.
Change in Gastrointestinal Angiodysplasia (GIAD) Foci | From Baseline to 180 days
  Microvascular angiodysplasia will be assessed by video capsule endoscopy (VCE). VCE is a minimally invasive technique used to identify gastrointestinal lesions and diagnose GIAD. Change in the group mean number of GIAD foci/lesions per patient from baseline to 180 days will be determined.
  GIAD formation will only be assessed at baseline and at 180 days unless the patient(s) experiences an episode of gastrointestinal bleeding prior to 180 days.
Change in Vascular Reactivity Index | From Baseline to 180 days
  Endothelial function will be determined by the finger vascular reactivity index (VRI) during LVAD support. VRI will be assessed by a non-invasive method using the Endothelix device. VRI is determined by measuring fingertip temperature change before and after cuff deflation. Change in group median VRI values from baseline will be summarized. Positive changes from baseline are associated with improved endothelial function.

SECONDARY OUTCOMES:
Change in Urinary Protein to Creatinine Ratio (PCR) | From Baseline to 180 days and, as available, 12, 18, and 24 months
  Urine samples will be assessed to determine the protein to creatinine ratio. Urinary PCR is calculated by dividing the concentration of protein (mg/dL) in the urine sample by the creatinine concentration (mg/dL). Change in group mean urinary protein to creatine ratios from baseline will be summarized. Elevated ratios of protein to creatinine are associated with increased risk of renal disease and microvascular dysfunction.
Platelet Gene Expression | Baseline, 3 months, and 6 months
  Platelet samples will be assessed for changes in gene expression using RNA sequencing analysis. Platelets will be isolated from whole blood samples collected at baseline, 3 months, and 6 months from participants in each group. Equal number of isolated platelets will be lysed in Trizol and DNAse treated total RNA will be isolated. RNA sequencing will be performed using HiSeq 50 Cycle Single Read Sequencing after library preparation. Differentially expressed genes (DEGs) will be ranked by their expression change between groups. DEGs with > 1.5-fold change in expression after LVAD at a sequence depth of >30 million reads per sample will be ranked by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Saeed, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL. Epidemiology of Heart Failure: A Contemporary Perspective. Circ Res. 2021 May 14;128(10):1421-1434. doi: 10.1161/CIRCRESAHA.121.318172. Epub 2021 May 13. PMID 33983838
- [Background] Molina EJ, Shah P, Kiernan MS, Cornwell WK 3rd, Copeland H, Takeda K, Fernandez FG, Badhwar V, Habib RH, Jacobs JP, Koehl D, Kirklin JK, Pagani FD, Cowger JA. The Society of Thoracic Surgeons Intermacs 2020 Annual Report. Ann Thorac Surg. 2021 Mar;111(3):778-792. doi: 10.1016/j.athoracsur.2020.12.038. Epub 2021 Jan 16. PMID 33465365
- [Background] Colombo PC, Mehra MR, Goldstein DJ, Estep JD, Salerno C, Jorde UP, Cowger JA, Cleveland JC Jr, Uriel N, Sayer G, Skipper ER, Downey FX, Ono M, Hooker R Jr, Anyanwu AC, Givertz MM, Mahr C, Topuria I, Somo SI, Crandall DL, Horstmanshof DA. Comprehensive Analysis of Stroke in the Long-Term Cohort of the MOMENTUM 3 Study. Circulation. 2019 Jan 8;139(2):155-168. doi: 10.1161/CIRCULATIONAHA.118.037231. PMID 30586698
- [Background] Yuzefpolskaya M, Schroeder SE, Houston BA, Robinson MR, Gosev I, Reyentovich A, Koehl D, Cantor R, Jorde UP, Kirklin JK, Pagani FD, D'Alessandro DA. The Society of Thoracic Surgeons Intermacs 2022 Annual Report: Focus on the 2018 Heart Transplant Allocation System. Ann Thorac Surg. 2023 Feb;115(2):311-327. doi: 10.1016/j.athoracsur.2022.11.023. Epub 2022 Dec 1. PMID 36462544
- [Background] Jorde UP, Saeed O, Koehl D, Morris AA, Wood KL, Meyer DM, Cantor R, Jacobs JP, Kirklin JK, Pagani FD, Vega JD. The Society of Thoracic Surgeons Intermacs 2023 Annual Report: Focus on Magnetically Levitated Devices. Ann Thorac Surg. 2024 Jan;117(1):33-44. doi: 10.1016/j.athoracsur.2023.11.004. Epub 2023 Nov 8. PMID 37944655
- [Background] Schmitto JD, Shaw S, Garbade J, Gustafsson F, Morshuis M, Zimpfer D, Lavee J, Pya Y, Berchtold-Herz M, Wang A, Gazzola C, Potapov E, Saeed D. Fully magnetically centrifugal left ventricular assist device and long-term outcomes: the ELEVATE registry. Eur Heart J. 2024 Feb 21;45(8):613-625. doi: 10.1093/eurheartj/ehad658. PMID 38036414
- [Background] Demirozu ZT, Radovancevic R, Hochman LF, Gregoric ID, Letsou GV, Kar B, Bogaev RC, Frazier OH. Arteriovenous malformation and gastrointestinal bleeding in patients with the HeartMate II left ventricular assist device. J Heart Lung Transplant. 2011 Aug;30(8):849-53. doi: 10.1016/j.healun.2011.03.008. Epub 2011 Apr 29. PMID 21530318
- [Background] Mattace-Raso FU, van der Cammen TJ, Hofman A, van Popele NM, Bos ML, Schalekamp MA, Asmar R, Reneman RS, Hoeks AP, Breteler MM, Witteman JC. Arterial stiffness and risk of coronary heart disease and stroke: the Rotterdam Study. Circulation. 2006 Feb 7;113(5):657-63. doi: 10.1161/CIRCULATIONAHA.105.555235. PMID 16461838
- [Background] Zieman SJ, Melenovsky V, Kass DA. Mechanisms, pathophysiology, and therapy of arterial stiffness. Arterioscler Thromb Vasc Biol. 2005 May;25(5):932-43. doi: 10.1161/01.ATV.0000160548.78317.29. Epub 2005 Feb 24. PMID 15731494
- [Background] Ambardekar AV, Hunter KS, Babu AN, Tuder RM, Dodson RB, Lindenfeld J. Changes in Aortic Wall Structure, Composition, and Stiffness With Continuous-Flow Left Ventricular Assist Devices: A Pilot Study. Circ Heart Fail. 2015 Sep;8(5):944-52. doi: 10.1161/CIRCHEARTFAILURE.114.001955. Epub 2015 Jul 1. PMID 26136459
- [Background] Ambardekar AV, Stratton MS, Dobrinskikh E, Hunter KS, Tatman PD, Lemieux ME, Cleveland JC, Tuder RM, Weiser-Evans MCM, Moulton KS, McKinsey TA. Matrix-Degrading Enzyme Expression and Aortic Fibrosis During Continuous-Flow Left Ventricular Mechanical Support. J Am Coll Cardiol. 2021 Nov 2;78(18):1782-1795. doi: 10.1016/j.jacc.2021.08.047. PMID 34711337
- [Background] Templeton DL, John R, Painter P, Kelly AS, Dengel DR. Effects of the left ventricular assist device on the compliance and distensibility of the carotid artery. Heart Vessels. 2013 May;28(3):377-84. doi: 10.1007/s00380-012-0271-4. Epub 2012 Aug 9. PMID 22875409
- [Background] Kiyatkin M, Stöhr E, Zuver A, Gaudig A, Yuzefpolskaya M, Colombo P and Willey J. Carotid artery flow and its assciation with stroke during left ventricular assist device support. Critical Care Medicine. 2019;47:53.
- [Background] Hackam DG, Spence JD. Antiplatelet Therapy in Ischemic Stroke and Transient Ischemic Attack. Stroke. 2019 Mar;50(3):773-778. doi: 10.1161/STROKEAHA.118.023954. No abstract available. PMID 30626286
- [Background] Lebas H, Yahiaoui K, Martos R, Boulaftali Y. Platelets Are at the Nexus of Vascular Diseases. Front Cardiovasc Med. 2019 Sep 11;6:132. doi: 10.3389/fcvm.2019.00132. eCollection 2019. PMID 31572732
- [Background] de Biasi AR, Manning KB, Salemi A. Science for surgeons: understanding pump thrombogenesis in continuous-flow left ventricular assist devices. J Thorac Cardiovasc Surg. 2015 Mar;149(3):667-73. doi: 10.1016/j.jtcvs.2014.11.041. Epub 2014 Nov 21. No abstract available. PMID 25534307
- [Background] Diehl P, Aleker M, Helbing T, Sossong V, Beyersdorf F, Olschewski M, Bode C, Moser M. Enhanced microparticles in ventricular assist device patients predict platelet, leukocyte and endothelial cell activation. Interact Cardiovasc Thorac Surg. 2010 Aug;11(2):133-7. doi: 10.1510/icvts.2010.232603. Epub 2010 May 14. PMID 20472650
- [Background] Liesdek OCD, Schutgens REG, de Heer LM, Ramjankhan FZ, Sebastian SAE, Rohof JJ, Suyker WJL, Urbanus RT. Acquired blood platelet disorder in patients with end-stage heart failure after implantation of a continuous centrifugal-flow left ventricular assist device: A prospective cohort study. Res Pract Thromb Haemost. 2023 Mar 6;7(2):100101. doi: 10.1016/j.rpth.2023.100101. eCollection 2023 Feb. PMID 37063754
- [Background] Radovancevic R, Matijevic N, Bracey AW, Radovancevic B, Elayda M, Gregoric ID, Frazier OH. Increased leukocyte-platelet interactions during circulatory support with left ventricular assist devices. ASAIO J. 2009 Sep-Oct;55(5):459-64. doi: 10.1097/MAT.0b013e3181b235af. PMID 19730003
- [Background] Griesshammer M, Beneke H, Nussbaumer B, Grunewald M, Bangerter M, Bergmann L. Increased platelet surface expression of P-selectin and thrombospondin as markers of platelet activation in essential thrombocythaemia. Thromb Res. 1999 Nov 1;96(3):191-6. doi: 10.1016/s0049-3848(99)00095-x. PMID 10588461